CLINICAL TRIAL: NCT00550927
Title: A Phase 1 Safety Evaluation of Oral Enzastaurin in Combination With Bevacizumab in Patients With Advanced/Metastatic Cancer
Brief Title: Enzastaurin and Bevacizumab in Treating Patients With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 11182; JHOC-J0688; JHOC-NA_00004943; CDR0000571514; H6Q-MC-S029 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-22; First posted 2007-10-30 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bevacizumab

INTERVENTIONS:
Biological: bevacizumab
Drug: enzastaurin hydrochloride
Other: diagnostic laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Enzastaurin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Enzastaurin and bevacizumab may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving enzastaurin together with bevacizumab may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of enzastaurin and bevacizumab in treating patients with locally advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the recommended phase II doses of enzastaurin hydrochloride and bevacizumab that may be safely administered to patients with locally advanced or metastatic malignancies.
* To characterize the toxicities of enzastaurin hydrochloride and bevacizumab in these patients.
* To document the antitumor activity of enzastaurin hydrochloride and bevacizumab in these patients.
* To evaluate the pharmacokinetics of enzastaurin hydrochloride and bevacizumab in these patients.
* To assess GSK3β as a biomarker relevant to enzastaurin hydrochloride and its correlation with clinical outcome in these patients.

OUTLINE: This is a dose-escalation study of enzastaurin hydrochloride and bevacizumab.

Patients receive oral enzastaurin hydrochloride once, twice, or three times daily on days 1-21 or days 1-28 and bevacizumab IV over 30-90 minutes on day 1 or days 1 and 15. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically during study for pharmacokinetic evaluation. Samples are also analyzed for biomarker (GSK3β) by ELISA.

After completion of study treatment, patients are followed for 30 days.

National Cancer Institute (NCI) registered this trial with Eli Lilly as sponsor. NCI did not update the record. In June 2012, NCI transferred the trial to Lilly's clinicaltrials.gov account and Lilly updated the record with the trial status and trial completion dates. This trial is not an applicable trial under Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic diagnosis of locally advanced or metastatic cancer for which no preferable therapy exists
* Measurable or nonmeasurable disease
* No CNS metastases or a primary CNS tumor

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* WBC count ≥ 3.0 × 10^9/L
* Absolute neutrophil count ≥ 1.5 × 10^9/L
* Platelet count ≥ 100 × 10^9/L
* Hemoglobin ≥ 10 g/dL (6.21 mmol/L)
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN (5 times ULN if liver metastases are present)
* AST and ALT ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Serum creatinine < 1.5 times ULN
* No proteinuria at baseline, as demonstrated by either of the following:

  * Urine protein:creatinine ratio < 1.0 at screening
  * Urine dipstick for proteinuria < 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline must undergo a 24-hour urine collection that demonstrates ≤ 1 g of protein in 24 hours to be eligible for study participation)
* No second primary malignancy that could affect compliance with the study or interpretation of the study results
* No concurrent serious systemic disorder (e.g., active infection, including HIV) that, in the opinion of the investigator, would compromise the patient's ability to adhere to the study
* No known hypersensitivity to bevacizumab or enzastaurin hydrochloride, or to a component of either drug
* No prior bevacizumab-related toxicity requiring discontinuation, such as a thromboembolic event, hemorrhage, or serious hypertension
* No clinically significant cardiac disease, in the opinion of the investigator, including any of the following:

  * Myocardial infarction within the past 6 months
  * Symptomatic angina pectoris
  * Congestive heart failure not controlled by medications
  * ECG abnormalities indicative of clinically significant cardiac disease
* No evidence of bleeding diathesis or coagulopathy
* No nonhealing cutaneous wound or gastrointestinal ulcer
* No history of or risk for abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No hemoptysis requiring medical attention within the past 3 months
* No known history of cerebrovascular accidents or transient ischemic attacks
* No clinically significant vascular or peripheral vascular disease
* No hypertension not controlled by medical management
* No history of hypertensive crisis or hypertensive encephalopathy
* No significant traumatic injury within the past 28 days
* Able to comply with study or study procedures
* Able to swallow tablets
* Exhibits compliance and geographic proximity that allow adequate follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* No prior participation in this study or any other study involving enzastaurin hydrochloride
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* At least 4 weeks since prior radiotherapy, anticancer hormone therapy, or other investigational therapy

  * Patients with hormone-refractory prostate cancer receiving luteinizing hormone-releasing hormone analogue therapy (leuprolide or goserelin) prior to study enrollment should continue therapy during study participation
* At least 6 weeks since prior bicalutamide
* At least 4 weeks since prior flutamide or nilutamide
* More than 10 days since prior and no concurrent aspirin > 325 mg/day
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior core biopsy or other minor surgical procedure, excluding placement of a vascular access device
* No concurrent carbamazepine, phenobarbital, or phenytoin
* No concurrent systemic anticoagulation
* No concurrent chronic use of other nonsteroidal anti-inflammatory drugs
* No concurrent routine use of colony-stimulating factors
* No concurrent major surgery
* No other concurrent chemotherapy, radiotherapy, immunotherapy, or experimental medications
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II doses of enzastaurin hydrochloride and bevacizumab
Safety
Time to disease progression
Overall response rate (complete and partial response)
Duration of response
Duration of stable disease
ECOG performance status over time
Pharmacokinetics
Biomarker (GSK3β) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Connie Collins, BSN — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Nwankwo N, Zhang Z, Wang T, Collins C, Resta L, Ermisch S, Day J, Decker R, Kornberg L, Nicol S, Thornton D, Armstrong DK, Carducci MA. Phase I study of enzastaurin and bevacizumab in patients with advanced cancer: safety, efficacy and pharmacokinetics. Invest New Drugs. 2013 Jun;31(3):653-60. doi: 10.1007/s10637-012-9850-6. Epub 2012 Jul 6. PMID 22766773